CLINICAL TRIAL: NCT06801977
Title: Genetic Susceptibility Study of Primary Pulmonary Lymphoepithelioma-like Carcinoma
Brief Title: The Chinese Pulmonary Lymphoepithelioma-like Carcinoma Collaboration Study
Acronym: CPLCC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Jia wei-hua, Professor, Sun Yat-sen University
Other Study IDs: SL-B2025-059-01
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Primary Pulmonary Lymphoepithelioma-like Carcinoma
Keywords: Genome-Wide Association Study; primary Pulmonary Lymphoepithelioma-like Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SYSUCC cohort, Guangdong, China: Cases:
  Patients aged 18 and above with a pathological diagnosis of primary pulmonary lymphoepithelioma-like carcinoma who were treated at the Sun Yat-sen University Cancer Center from January 1, 2002.
  Controls:
  Healthy participants aged 18 and above.
  Interventions: Genetic: Genome-wide genotyping
- Foshan cohort, Guangdong, China: Cases:
  Patients aged 18 and above with a pathological diagnosis of primary pulmonary lymphoepithelioma-like carcinoma who were treated at the the First People's Hospital of Foshan from January 1, 2007.
  Controls:
  Healthy participants aged 18 and above.
  Interventions: Genetic: Genome-wide genotyping

INTERVENTIONS:
Genetic: Genome-wide genotyping — Whole blood from the participants was used to extract DNA for genotyping.

SUMMARY:
This retrospective case-control study aims to investigate the genetic mechanisms of primary Pulmonary Lymphoepithelioma-like Carcinoma, identify genetic susceptibility loci associated with its onset, and explore potential pathogenic genes, providing new insights for its etiological research.

DETAILED DESCRIPTION:
Pulmonary lymphoepithelioma-like carcinoma (pLELC) is a rare non-small cell lung cancer (NSCLC) that histologically resembles nasopharyngeal carcinoma (NPC) and predominantly affects the Asian population. Epstein-Barr virus (EBV) infection is a recognized pathogenic factor, and the regional prevalence of pLELC suggests that genetic susceptibility also plays an important role. However, no genetic studies on pLELC have been conducted, leaving its genetic etiology poorly understood. In this study, genotyping for all the subjects was performed by using Illumina Infinium Global Screening Array. Genome-wide association followed by meta-analysis was performed for pLELC cases and healthy controls. The primary objective of this study is to discover susceptibility genes that explain the genetic mechanisms of pLELC.

ELIGIBILITY:
Case:

Inclusion criteria:

The subject is pathologically diagnosed with primary pulmonary lymphoepithelioma-like carcinoma.

Exclusion criteria:

The subject is diagnosed with metastatic nasopharyngeal carcinoma; The subject has heavy cardiovascular, liver, or kidney disease.

Controls:

Inclusion criteria:

The subject is in good physical condition and has a stable level of consciousness;

Exclusion criteria:

The subject has prevalent cancer; The subject has heavy cardiovascular, liver, or kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of cases and controls with specific inclusion and exclusion criteria. Cases were individuals pathologically diagnosed with primary pulmonary lymphoepithelioma-like carcinoma (PLELC), excluding those with metastatic nasopharyngeal carcinoma or severe cardiovascular, liver, or kidney disease. Controls were individuals in good physical condition with stable levels of consciousness, excluding those with a history of cancer or severe cardiovascular, liver, or kidney disease.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2002-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the occurrence of Pulmonary Lymphoepithelioma-like Carcinoma | The enrollment of the participants
  pathological diagnosis of Pulmonary Lymphoepithelioma-like Carcinoma

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Foshan First People's Hospital, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
To prioritize participant confidentiality and privacy, we have decided not to release Individual Participant Data (IPD). This decision reflects our commitment to safeguarding the sensitive information of participants, in full compliance with ethical standards and privacy laws. It is taken to protect the well-being and privacy of all individuals involved in the study.